CLINICAL TRIAL: NCT02329535
Title: Comparing a Double Dose of Vaginal Progesterone to no Treatment for the Prevention of Preterm Birth in Twins Pregnancy and Short Cervix
Brief Title: Comparing Double Dose of Vaginal Progesterone to no Treatment for Prevention of Preterm Birth in Twins and Short Cervix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results from similar research were already published
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Noah Zafran, Senion physician OB-GYN, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMC-005413-CTIL
Record Dates: First submitted 2014-11-30; First posted 2014-12-31 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Treatment with 400 mg Micronized progesterone (Utrogestan) daily up to 6 weeks of geastation
  Interventions: Drug: Micronized progesterone
- No treatment (No Intervention): No treatment. Regular follow up

INTERVENTIONS:
Drug: Micronized progesterone — vaginal caps 400 mg daily up to 36 weeks of gestation
  Other Names: Utrogestan
  Arms: Treatment group

SUMMARY:
Twin pregnancies are more likely to be delivered preterm than singleton pregnancies. Vaginal progesterone administration (200 mg Utrogestan) to asymptomatic women with a singleton pregnancy and sonographic short cervix reduced the risk of preterm birth (PTB) and neonatal morbidity and mortality, yet not proved efficient in twins' pregnancy. The investigators' hypothesis is that a higher dose of vaginal micronized progesterone will be more effective in preventing PTD. The objectives of the study is to compare the rate of preterm birth and perinatal morbidity and mortality in a twin pregnancy with short cervical length treated with vaginal 400 mg of micronized progesterone to no treatment. The study is Randomized, open label, of twin pregnancy between 16-26 weeks of gestation with cervical length under 25 mm. Women will be randomly assigned to either treatment or no treatment group. Progesterone treatment will be given until 36 weeks of gestation. Other management will be according to standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* Twin gestation
* Certain dating (documented first trimester ultrasound, or a reliable menstrual date confirmed by an ultrasound performed before 20 weeks of gestation)
* Age > 18 years
* Gestational age 16-26
* Cervical length<25 mm
* Intact membranes
* Informed consent

Exclusion Criteria:

* Major malformation or chromosomal abnormality to at least one fetus
* Higher order pregnancy
* Mocochorional-monoamniotic twin
* Death of one fetus
* Cervical dilatation >3 cm
* Chronic medical conditions that would interfere with study participation or evaluation of the treatment (e.g. seizures, psychiatric disorders, uncontrolled chronic hypertension, congestive heart failure, chronic renal failure, uncontrolled diabetes mellitus with end-organ dysfunction, active thrombophlebitis or a thromboembolic disorder, history of hormone-associated thrombophlebitis or thromboembolic disorders, active liver dysfunction or disease, known or suspected malignancy of the breast or genital organs)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Preterm delivery | up to 25 weeks from randomization
  Rate of preterm delivery before 37.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Head of delivery room, Department of OB-GYN, Emek medical center, Afula, Israel
Locations (2):
- Israel (2):
  - Haemek Medical Center, Afula
  - The Nazareth hospital, Nazareth

REFERENCES:
- [Background] Vayssiere C, Favre R, Audibert F, Chauvet MP, Gaucherand P, Tardif D, Grange G, Novoa A, Descamps P, Perdu M, Andrini E, Janse-Marec J, Maillard F, Nisand I. Cervical length and funneling at 22 and 27 weeks to predict spontaneous birth before 32 weeks in twin pregnancies: a French prospective multicenter study. Am J Obstet Gynecol. 2002 Dec;187(6):1596-604. doi: 10.1067/mob.2002.127380. PMID 12501070
- [Background] Skentou C, Souka AP, To MS, Liao AW, Nicolaides KH. Prediction of preterm delivery in twins by cervical assessment at 23 weeks. Ultrasound Obstet Gynecol. 2001 Jan;17(1):7-10. doi: 10.1046/j.1469-0705.2001.00357.x. PMID 11244660
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] DeFranco EA, O'Brien JM, Adair CD, Lewis DF, Hall DR, Fusey S, Soma-Pillay P, Porter K, How H, Schakis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Vaginal progesterone is associated with a decrease in risk for early preterm birth and improved neonatal outcome in women with a short cervix: a secondary analysis from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):697-705. doi: 10.1002/uog.5159. PMID 17899571
- [Background] Serra V, Perales A, Meseguer J, Parrilla JJ, Lara C, Bellver J, Grifol R, Alcover I, Sala M, Martinez-Escoriza JC, Pellicer A. Increased doses of vaginal progesterone for the prevention of preterm birth in twin pregnancies: a randomised controlled double-blind multicentre trial. BJOG. 2013 Jan;120(1):50-7. doi: 10.1111/j.1471-0528.2012.03448.x. Epub 2012 Aug 13. PMID 22882759
- [Background] Senat MV, Porcher R, Winer N, Vayssiere C, Deruelle P, Capelle M, Bretelle F, Perrotin F, Laurent Y, Connan L, Langer B, Mantel A, Azimi S, Rozenberg P; Groupe de Recherche en Obstetrique et Gynecologie. Prevention of preterm delivery by 17 alpha-hydroxyprogesterone caproate in asymptomatic twin pregnancies with a short cervix: a randomized controlled trial. Am J Obstet Gynecol. 2013 Mar;208(3):194.e1-8. doi: 10.1016/j.ajog.2013.01.032. PMID 23433324
- [Background] To MS, Fonseca EB, Molina FS, Cacho AM, Nicolaides KH. Maternal characteristics and cervical length in the prediction of spontaneous early preterm delivery in twins. Am J Obstet Gynecol. 2006 May;194(5):1360-5. doi: 10.1016/j.ajog.2005.11.001. Epub 2006 Apr 21. PMID 16647922
- [Background] Rode L, Klein K, Nicolaides KH, Krampl-Bettelheim E, Tabor A; PREDICT Group. Prevention of preterm delivery in twin gestations (PREDICT): a multicenter, randomized, placebo-controlled trial on the effect of vaginal micronized progesterone. Ultrasound Obstet Gynecol. 2011 Sep;38(3):272-80. doi: 10.1002/uog.9093. PMID 21739497